CLINICAL TRIAL: NCT01988558
Title: A Phase I/II, Randomized, Double Blind, Placebo-controlled Study to Assess the Safety, Tolerability and Efficacy of DL-lactic Acid Syrup (Tonsitin) in Children With Recurrent Tonsillitis.
Brief Title: A Phase I/II to Assess Safety, Tolerability and Efficacy of DL-lactic Acid Syrup in Children With Recurrent Tonsillitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yali Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LA-001-IL
Record Dates: First submitted 2013-11-03; First posted 2013-11-20 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Recurrent Tonsillitis in Children
Keywords: Recurrent Tonsillitis; Streptococcus A
MeSH Terms: conditions — Tonsillitis | interventions — Lactic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Treated Group (Experimental): Children diagnosed as suffering from recurrent Tonsillitis (at least 4 episodes per year) to receive DL-Lactic acid syrup twice a day for a month.
  Interventions: Drug: DL - Lactic Acid
- Placebo Group (Placebo Comparator)
  Interventions: Dietary Supplement: Raspberry flavored syrup

INTERVENTIONS:
Drug: DL - Lactic Acid — Treated group to receive DL - Lactic Acid Syrup (Raspberry flavored)
  Arms: Treated Group
Dietary Supplement: Raspberry flavored syrup — Placebo group to receive Raspberry flavored Syrup
  Arms: Placebo Group

SUMMARY:
The study objectives are to evaluate Tonsitin™ (10% Lactic Acid) safety, tolerability and preliminary efficacy, as a potent treatment for Recurrent Tonsillitis in children.

ELIGIBILITY:
Inclusion Criteria:

* Children at the ages of 5-16.
* Patient is suffering from recurrent documented sore throat with at least 4 tonsillitis episodes during the preceding year (at least one verified by culture or rapid antigen testing for Streptococcus A).
* Patient with clinical presentation of irregular tonsils.
* Tonsils size graded between 2.5-4.
* Clinical diagnosis of bacterial known in recurrent pharyngeal-tonsillitis.
* Patient is willing to participate in the study and adhere to the study protocol
* Patient's guardian and/or Patient have signed informed consent.

Exclusion Criteria:

* Clinical diagnosis of acute tonsillitis/pharyngitis caused by Streptococcus pyogenes (Positive RSAT or microbial culture).
* Subjects who are known as Streptococcus pyogenes carriers
* Subject's requiring any other medication (topical or systemic) that may affect the course of the disease during the study period (e.g. antibiotics, sedating antihistamines), and/or did not completed 14 days from end of antibiotics treatment.
* Subjects with known hypersensitivity to lactose.
* Subject is suffering from peritonsillar abscess.
* Subject suffers from an active peptic ulcer
* Subjects who are suffering from any concomitant disease which in the judgment of the investigator will interfere with the conduct or interpretation of the study results.
* Subject is currently participating in another clinical study.

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2013-12; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Safety evaluation - Number of participants with adverse events | At 90 days post treatment

SECONDARY OUTCOMES:
Tonsil Size | Chnge from baseline at 6 months post treatment
Number of Tonsillitis episodes | Chnge in medical history number of recurrent Tonsillitis episodes within 6 months post treatment

OTHER OUTCOMES:
QOL Questionnaire | Chnge from baseline at 90 days post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mati Berkovitz, Prof., Principal Investigator — MOH
Locations (3):
- Israel (3):
  - Clalit Health Services, Pediatric Community Ambulatory Clinic, Petah Tikva, Israel
  - Clalit Health Services, Pediatric Community Ambulatory Ganei Hadar clinic, Petah Tikva, Israel
  - Assaf Harofeh Medical Center, Tzrifin